CLINICAL TRIAL: NCT00775450
Title: Safety and Immunogenicity of Revaccination With Influenza Vaccine in Ambulatory Elderly Subjects Previously Vaccinated With Fluzone ID, Fluzone HD, and Fluzone® IM
Brief Title: Influenza Vaccine Revaccination in Ambulatory Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FID21
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Influenza; Orthomyxovirus Infection; Myxovirus Infection
Keywords: Influenza; Orthomyxovirus Infection; Inactivated Split-virion influenza vaccine; Elderly
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1a: Fluzone ID After Fluzone ID (Experimental)
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 1b: Fluzone IM After Fluzone ID (Experimental)
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 2a: Fluzone IM After Fluzone IM (Active Comparator)
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 2b: Fluzone ID After Fluzone IM (Experimental)
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 3: Fluzone HD After Fluzone HD (Active Comparator)
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B

INTERVENTIONS:
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Other Names: Fluzone
  Arms: Group 1a: Fluzone ID After Fluzone ID
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.5 mL, Intramuscular
  Other Names: Fluzone
  Arms: Group 1b: Fluzone IM After Fluzone ID
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.5 mL, Intramuscular
  Other Names: Fluzone
  Arms: Group 2a: Fluzone IM After Fluzone IM
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Other Names: Fluzone
  Arms: Group 2b: Fluzone ID After Fluzone IM
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.5 mL, Intramuscular
  Other Names: Fluzone
  Arms: Group 3: Fluzone HD After Fluzone HD

SUMMARY:
This is a multi-center study designed to evaluate the safety and immunogenicity of a Fluzone revaccination in elderly adults aged ≥ 65 years.

Primary Objective:

To describe the safety profile for all subjects.

Secondary Objective:

To describe immunogenicity 28 days following revaccination with one of three Fluzone formulations.

DETAILED DESCRIPTION:
Subjects who previously participated in study FID29 will be invited to participate in this revaccination study. They will be assigned to 1 of 3 groups based on the group they were previously randomized to and the vaccine received in study FID29.

ELIGIBILITY:
Inclusion Criteria :

* Aged ≥ 65 years on the day of vaccination
* Enrolled in and completed study FID29 and received the correct vaccine for the group to which they were randomized
* Informed consent form signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* Subject is medically stable.

Exclusion Criteria :

* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the four weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccination in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Known human immunodeficiency virus (HIV), hepatitis B (HBs) antigen, or Hepatitis C seropositivity.
* Previous vaccination against influenza in the past 6 months with the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular (IM) vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Neoplastic disease or any hematologic malignancy, (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, as well as subjects who have a history of neoplastic disease and who have been disease free for ≥ 5 years).
* Personal or family history of Guillain-Barré Syndrome.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 807 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (27):
- United States (27):
  - Hoover, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fountain Valley, California
  - San Diego, California
  - Milford, Connecticut
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Chicago, Illinois
  - Wichita, Kansas
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Fort Worth, Texas
  - Galveston, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Marshfield, Wisconsin

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 October to 20 November 2008 in 27 medical centers in the US.
Pre-assignment Details: A total of 807 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1a: Fluzone ID After Fluzone ID: Participants who received a dose (0.1 mL) of Fluzone intradermal (ID) after receiving Fluzone ID in Study FID29 (NCT00551031)
- Group 1b: Fluzone IM After Fluzone ID: Participants who received a dose (0.5 mL) of Fluzone intramuscular (IM) vaccine after receiving Fluzone intradermal (ID) vaccine in Study FID29 (NCT00551031)
- Group 2a: Fluzone IM After Fluzone IM: Participants who received a dose (0.5 mL) Fluzone intramuscular (IM) vaccine after receiving Fluzone IM vaccine in Study FID29 NCT00551031)
- Group 2b: Fluzone ID After Fluzone IM: Participants who received a dose (0.1 )Fluzone intradermal (ID) vaccine after receiving Fluzone intramuscular (IM) vaccine in Study FID29 (NCT00551031)
- Group 3: Fluzone HD After Fluzone HD: Participants who received a dose (0.5 mL) of Fluzone High Dose (HD) vaccine after receiving Fluzone HD vaccine in Study FID29 (NCT00551031)
Period: Overall Study
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD
Started | 295 | 98 | 105 | 108 | 201
Completed | 292 | 98 | 105 | 108 | 199
Not Completed | 3 | 0 | 0 | 0 | 2
Not completed — Serious Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD | Total
Number analyzed (Participants) | 295 | 98 | 105 | 108 | 201 | 807
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 295 | 98 | 105 | 108 | 201 | 807
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.9 (5.99) | 74.2 (5.97) | 73.0 (5.37) | 74.3 (5.11) | 73.5 (5.74) | 73.8 (5.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 54 | 58 | 61 | 117 | 459
  Male | 126 | 44 | 47 | 47 | 84 | 348
Region of Enrollment [Number; unit: participants]
  United States | 295 | 98 | 105 | 108 | 201 | 807

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions After Fluzone Intradermal or Fluzone Intramuscular or Fluzone High-dose Vaccine Injection
Description: Solicited injection site reactions: Pain, Erythema (redness), Swelling, Induration, Ecchymosis, Pruritus. Solicited systemic reactions: Fever, (Temperature), Headache, Malaise, Myalgia, and Shivering.
Time Frame: Days 0 through 7 post vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD
Number analyzed (Participants) | 292 | 98 | 105 | 107 | 200
Participants
  Any Solicited Injection site Pain | 68 | 18 | 23 | 31 | 91
  Grade 3 Pain (Incapacitating) | 2 | 0 | 0 | 2 | 1
  Any Solicited Injection site Erythema | 207 | 18 | 9 | 71 | 34
  Grade 3 Erythema (≥ 5 cm) | 34 | 1 | 0 | 7 | 7
  Any Solicited Injection site Swelling | 127 | 4 | 3 | 44 | 23
  Grade 3 Swelling (≥ 5 cm) | 9 | 0 | 0 | 3 | 5
  Any Solicited Injection site Induration | 133 | 6 | 6 | 50 | 18
  Grade 3 Induration (≥ 5 cm) | 5 | 0 | 0 | 1 | 1
  Any Solicited Injection site Ecchymosis | 27 | 2 | 5 | 11 | 6
  Grade 3 Ecchymosis (≥ 5 cm) | 1 | 0 | 0 | 0 | 0
  Any Solicited Injection site Pruritus | 99 | 3 | 6 | 38 | 20
  Grade 3 Pruritus (Incapacitating) | 6 | 0 | 0 | 1 | 0
  Any Fever | 9 | 1 | 1 | 4 | 7
  Grade 3 Fever (>102.2 ºF) | 0 | 0 | 0 | 0 | 0
  Any Headache | 39 | 14 | 15 | 17 | 45
  Grade 3 Headache (Prevents daily activities) | 1 | 0 | 0 | 2 | 1
  Any Malaise | 31 | 7 | 18 | 16 | 36
  Grade 3 Malaise (Prevents daily activities) | 1 | 0 | 0 | 1 | 2
  Any Myalgia | 35 | 18 | 25 | 22 | 48
  Grade 3 Myalgia (Prevents daily activities) | 0 | 0 | 0 | 1 | 2
  Any Shivering | 12 | 2 | 5 | 7 | 9
  Grade 3 Shivering (Prevents daily activities) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Geometric Mean Titers (GMTs) Before and After Vaccination With Fluzone Intradermal or Fluzone Intramuscular or Fluzone High-dose Vaccine Injection
Description: Serum antibody titers for the influenza vaccine serogroups A/H1N1, A/H3N2, and B were assessed by the hemagglutinin inhibition (HAI) assay.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Serum antibody titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD
Number analyzed (Participants) | 273 | 94 | 100 | 102 | 187
Titers
  A/H1N1 Pre-dose (Day 0,N = 273, 94, 100, 102, 186) | 28.7 [25.3 to 32.5] | 23.5 [19.3 to 28.6] | 27.3 [22.0 to 33.9] | 20.8 [17.1 to 25.2] | 28.7 [24.5 to 33.6]
  A/H1N1 Post -dose (Day 0 = 273, 94, 100, 102, 185) | 75.0 [66.4 to 84.7] | 59.6 [48.4 to 73.2] | 72.4 [58.7 to 89.2] | 73.5 [60.4 to 89.5] | 113 [96.2 to 133]
  A/H2N3 Pre-dose (Day 0, N= 273, 94, 100, 102, 186) | 30.8 [26.3 to 36.2] | 28.7 [22.1 to 37.3] | 24.5 [19.6 to 30.7] | 28.1 [21.8 to 36.2] | 36.6 [30.2 to 44.4]
  A/H2N3 Post Dose (n = 273, 94, 100, 102, 187) | 244 [205 to 289] | 212 [156 to 288] | 257 [197 to 336] | 273 [208 to 358] | 454 [380 to 543]
  B Pre Dose (n = 273, 94, 100, 102, 186 | 22.8 [20.2 to 25.6] | 18.9 [15.5 to 22.9] | 21.8 [18.0 to 26.5] | 21.9 [17.9 to 26.8] | 22.3 [19.6 to 25.4]
  B Post Dose (n = 273, 94, 100, 102, 185) | 54.3 [48.3 to 61.0] | 51.4 [42.4 to 62.3] | 60.4 [49.6 to 73.6] | 51.1 [42.9 to 60.9] | 78.2 [68.5 to 89.3]

3. Secondary Outcome: Percentage of Participants Who Achieved Seroprotection Post-Vaccination With Fluzone Intradermal or Fluzone Intramuscular or Fluzone High-dose Vaccine
Description: Seroprotection was defined as hemagglutinin inhibition (HAI) titer ≥ 1:40 at Day 28.
Time Frame: Days 0 and 28 post-vaccination
Population: Serum antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD
Number analyzed (Participants) | 273 | 94 | 100 | 102 | 187
Percentage of Participants
  A/H1N1 Serogroup - (Day 0, Pre-dose) | 40 | 36 | 39 | 26 | 41
  A/H1N1 Serogroup - (Day 28, Post-dose) | 80 | 72 | 80 | 81 | 88
  A/H3N2 Serogroup - (Day 0, Pre-dose) | 49 | 40 | 38 | 48 | 50
  A/H3N2 Serogroup - (Day 28, Post-dose) | 93 | 86 | 94 | 91 | 98
  B Serogroup - (Day 0, Pre-dose) | 36 | 29 | 32 | 32 | 36
  B Serogroup - (Day 28, Post-dose) | 73 | 69 | 75 | 66 | 83

4. Secondary Outcome: Percentage of Participants Who Achieved Seroconversion Post-Vaccination With Fluzone Intradermal or Fluzone Intramuscular or Fluzone High-dose Vaccine
Description: Seroconversion was defined as either a pre-vaccination hemagglutinin inhibition (HAI) titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre- vaccination titer ≥ 1:10 and a minimum 4 fold increase at 28 days post vaccination.
Time Frame: Day 28 post vaccination
Population: Serum antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD
Number analyzed (Participants) | 273 | 94 | 100 | 102 | 186
Percentage of Participants
  A/H1N1 (N = 273, 94, 100, 102, 185) | 31 | 28 | 31 | 44 | 47
  A/H2N3 (N = 273, 94, 100, 102, 186) | 73 | 64 | 76 | 75 | 84
  B (N = 273, 94, 100, 102, 185) | 24 | 31 | 33 | 26 | 41

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to up to 6 months post-vaccination
Arm/Group | Group 1a: Fluzone ID After Fluzone ID | Group 1b: Fluzone IM After Fluzone ID | Group 2a: Fluzone IM After Fluzone IM | Group 2b: Fluzone ID After Fluzone IM | Group 3: Fluzone HD After Fluzone HD
Serious Adverse Events (participants affected / at risk) | 10/295 | 3/98 | 6/105 | 3/108 | 10/201
Other Adverse Events (participants affected / at risk) | 239/292 | 42/98 | 54/105 | 86/107 | 123/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1a: Fluzone ID After Fluzone ID (N=295) | Group 1b: Fluzone IM After Fluzone ID (N=98) | Group 2a: Fluzone IM After Fluzone IM (N=105) | Group 2b: Fluzone ID After Fluzone IM (N=108) | Group 3: Fluzone HD After Fluzone HD (N=201)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Media Chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1a: Fluzone ID After Fluzone ID (N=292) | Group 1b: Fluzone IM After Fluzone ID (N=98) | Group 2a: Fluzone IM After Fluzone IM (N=105) | Group 2b: Fluzone ID After Fluzone IM (N=107) | Group 3: Fluzone HD After Fluzone HD (N=200)
Injection Site Pain (General disorders) | 68 (68) | 18 (18) | 23 (23) | 31 (31) | 91 (91)
Injection Site Erythema (General disorders) | 207 (207) | 18 (18) | 9 (9) | 71 (71) | 34 (34)
Injection Site Swelling (General disorders) | 127 (127) | 4 (4) | 3 (3) | 44 (44) | 23 (23)
Injection Site Induration (General disorders) | 133 (133) | 6 (6) | 6 (6) | 50 (50) | 18 (18)
Injection Site Ecchymosis (Vascular disorders) | 27 (27) | 2 (2) | 5 (5) | 11 (11) | 6 (6)
Injection Site Pruritus (Skin and subcutaneous tissue disorders) | 99 (99) | 3 (3) | 6 (6) | 38 (38) | 20 (20)
Malaise (General disorders) | 31 (31) | 7 (7) | 18 (18) | 16 (16) | 36 (36)
Shivering (General disorders) | 12 (12) | 2 (2) | 5 (5) | 7 (7) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (35) | 18 (18) | 25 (25) | 22 (22) | 48 (48)
Headache (Nervous system disorders) | 39 (39) | 14 (14) | 15 (15) | 17 (17) | 45 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.